CLINICAL TRIAL: NCT01419431
Title: Increased SOCS 3 mRNA in Monocytes From Patients Subjected to Laparoscopic Colon Surgery
Brief Title: Attenuated Inflammatory Response in Laparoscopic Colon Surgery
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Dag T Førland, MD, Oslo University Hospital
Other Study IDs: SOCS3 mRNA; SOCS-3-202008 (Other Grant/Funding Number: OUS-SOCS3)
Record Dates: First submitted 2011-07-18; First posted 2011-08-18 (Estimated); Last update posted 2011-12-16 (Estimated); Status verified 2011-12

CONDITIONS: Regulation of Inflammatory Response
Keywords: Colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colon cancer patients: Laparoscopic resection
  Interventions: Procedure: Laparoscopic resection

INTERVENTIONS:
Procedure: Laparoscopic resection — Inflammatory response in laparoscopic surgery
  Other Names: Colon cancer

SUMMARY:
Pro-inflammatory responses following laparoscopic surgery.

DETAILED DESCRIPTION:
Blood samples from 20 patient with colon cancer collected before and in 3 days following laparoscopic surgery. Analyzed for inflammatory cytokines and corresponding SOCS3 mRNA.

ELIGIBILITY:
Inclusion Criteria:Colon cancer stage I-III -

Exclusion Criteria:Colon cancer stage IV

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colon cancer stage I-III
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Inflammatory values for laparoscopic resection for colon cancer. | 3 days
  Corresponding values of SOCS3 mRNA copared to inflammatory cytokines in patients with laparoscopic resection for colon cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Dag T. Førland, MD, Principal Investigator — OUS
Locations (1):
- Oslo University Hospital, Oslo, Norway